CLINICAL TRIAL: NCT02132676
Title: Peer Support to Enhance Diabetes Shared Medical Appointments: Examining Comparative Effectiveness in VA Health Systems
Brief Title: Shared Health Appointments and Reciprocal Enhanced Support
Acronym: SHARES
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IIR 15-321
Record Dates: First submitted 2013-08-21; First posted 2014-05-07 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Insipidus
Keywords: Self-Management; Patient Care Management; Peer Group; Disease Management; Health Plan Implementation; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Insipidus; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Active treatment: All those scheduled for a Shared Medical Appointment (SMA), regardless of whether the Peer to Peer (P2P) program was offered.
- Usual Care: The randomly selected sample of those not offered participation in a Shared Medical Appointment (SMA).

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a peer-to-peer program (P2P) in addition to Shared Medical Appointments (SMAs) compared to SMAs alone for the treatment of diabetes in five VA health systems, and to study the implementation process in order to gather information required to disseminate the program more broadly in the VHA system.

DETAILED DESCRIPTION:
Providers are often unable to communicate as frequently as needed with diabetes patients who have poor risk factor control and face significant self-management challenges. Moreover, many VA patients face barriers to attending frequent face-to-face visits. This project will evaluate the implementation of a novel program found in a recent VA randomized, controlled trial to significantly improve VA patients' diabetes-specific social support, insulin starts, and glycemic control compared to usual nurse care management. The program uses periodic group sessions in conjunction with calls between paired patients with diabetes to promote more effective care management as well as peer-to-peer (P2P) communication among diabetes patients who both have poor glycemic control and are working on similar care goals. "Peer buddies" are encouraged to talk by phone at least weekly to provide mutual support and share their progress on meeting their self-management goals. The goal of this service is to enhance the effect of shared medical appointments (SMAs), a service model demonstrated to be effective in improving outcomes among patients with diabetes and other chronic conditions and now being widely implemented in VA. Based on the success of the efficacy trial of this intervention, the investigators now seek to evaluate a wider-scale implementation of this program. During implementation of the P2P program in conjunction with shared medical appointments (SMAs) in five diverse VA facilities, the investigators will evaluate the effectiveness of SMAs alone and SMAs+P2P compared to usual care, and study the implementation process in order to gather information required to disseminate the program more broadly in Veterans Health Administration (VHA).

ELIGIBILITY:
Inclusion Criteria:

Veterans enrolled into diabetes Shared Medical Appointments (SMAs) at participating sites, and a random subset of those meeting criteria for diabetes SMAs who have not yet participated:

* Veteran receiving care at a participating VA Medical Center
* Meets at least one of the following criteria in the past 2 years;

  * at least 1 VA hospitalization with a diabetes-related International Classification Of Diseases-9 (ICD-9) code,
  * at least 2 VA outpatient visits with a diabetes-related ICD-9 code, or
  * At least 1 VA prescription for a glucose control medication (insulin or oral agent) or monitoring supplies
* Poor glycemic control, indicated by a HbA1c in the past 6 months or:

  * at least 7.5% if age <70, or
  * at least 8% if age 70+
* Has a current address and telephone number listed in VA databases
* Is competent to provide informed consent
* Can communicate in English and by telephone
* Able to participate in an outpatient program

Exclusion Criteria:

For no intervention control group:

* Active substance abuse disorder (smoking cigarettes is not an exclusion)
* Serious psychiatric illness (bipolar disorder, dementia, schizophrenia, or personality disorders)
* Terminally ill
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: VA outpatients with uncontrolled diabetes receiving care at a participating VA Medical Center during implementation of a P2P program for diabetes management in conjunction with SMAs
Sampling Method: Non-Probability Sample
Enrollment: 1536 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ellen M Heisler, MD MPA, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (5):
- United States (5):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Northern California Health Care System, Mather, CA, Sacramento, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heisler M, Burgess J, Cass J, Chardos JF, Guirguis AB, Jeffery SM, Strohecker LA, Tremblay AS, Wu WC, Zulman DM. The Shared Health Appointments and Reciprocal Enhanced Support (SHARES) study: study protocol for a randomized trial. Trials. 2017 May 26;18(1):239. doi: 10.1186/s13063-017-1959-7. PMID 28549471
- [Background] Kowalski CP, Veeser M, Heisler M. Formative evaluation and adaptation of pre-and early implementation of diabetes shared medical appointments to maximize sustainability and adoption. BMC Fam Pract. 2018 Jul 7;19(1):109. doi: 10.1186/s12875-018-0797-3. PMID 29981568
- [Derived] Heisler M, Burgess J, Cass J, Chardos JF, Guirguis AB, Strohecker LA, Tremblay AS, Wu WC, Zulman DM. Evaluating the Effectiveness of Diabetes Shared Medical Appointments (SMAs) as Implemented in Five Veterans Affairs Health Systems: a Multi-site Cluster Randomized Pragmatic Trial. J Gen Intern Med. 2021 Jun;36(6):1648-1655. doi: 10.1007/s11606-020-06570-y. Epub 2021 Feb 2. PMID 33532956

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Randomly selected sample of those not offered participation in a Shared Medical Appointment (SMA)
- Active Treatment: All those scheduled for a Shared Medical Appointment (SMA), regardless of whether an SMA was actually attended
Period: Overall Study
Arm/Group | Usual Care | Active Treatment
Started | 727 | 809
Completed | 727 | 809
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Active Treatment | Total
Number analyzed (Participants) | 727 | 809 | 1536
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (12.7) | 67.1 (9.2) | 67.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 27 | 47
  Male | 707 | 782 | 1489
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 7 | 13
  Asian | 23 | 27 | 50
  Native Hawaiian or Other Pacific Islander | 9 | 14 | 23
  Black or African American | 85 | 148 | 233
  White | 536 | 545 | 1081
  More than one race | 7 | 8 | 15
  Unknown or Not Reported | 61 | 60 | 121
A1c [Mean (Standard Deviation); unit: percent] | 8.9 (1.3) | 9.1 (1.5) | 9.0 (1.4)
SBP [Mean (Standard Deviation); unit: mmHg] | 137.7 (15.2) | 136.2 (13.4) | 136.8 (14.2)
On insulin [Count of Participants; unit: Participants] | 255 | 385 | 640
On statin [Count of Participants; unit: Participants] | 470 | 603 | 1073
Classes of anti-hypertensive meds [Mean (Standard Deviation); unit: number of classes of antihypertensives] | 2.2 (1.3) | 2.4 (1.2) | 2.3 (1.2)
Primary Care Physician (PCP) in-person visits in past 8 months [Mean (Standard Deviation); unit: number of in-person PCP visits] | 3.2 (3.4) | 3.4 (3.1) | 3.3 (3.3)
PCP phone visits in past 8 months [Mean (Standard Deviation); unit: number of PCP phone visits] | 0.7 (1.5) | 0.7 (1.2) | 0.7 (1.3)
Nurse case manager in-person visits in past 8 months [Mean (Standard Deviation); unit: number of RNCM in-person visits] | 0.2 (0.8) | 0.2 (0.7) | 0.2 (0.7)
Nurse case manager phone visits in past 8 months [Mean (Standard Deviation); unit: number of RNCM phone visits] | 0.3 (0.9) | 0.3 (0.9) | 0.3 (0.9)
Endocrinology in-person visits in past 8 months [Mean (Standard Deviation); unit: number of Endocrinology in-person visits] | 0.2 (0.8) | 0.3 (0.8) | 0.3 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycemic Control
Description: Glycemic control (measured by Hemoglobin A1c) in each group will be assessed by the comparison of an average of the values obtained during routine outpatient clinical practice in 6-month windows preceding baseline and following the 6 and 12-month post-enrollment evaluation periods. In addition to measuring absolute values of A1c, the investigators will also examine the change in the percentage of patients with an average A1c > 8%.
Time Frame: 6 months and 12 months post-enrollment
Population: Only those with A1c values documented in the electronic health record (EHR) during the evaluation windows were included in the number analyzed
Measure: Mean (Standard Deviation); unit: % glycolated hemoglobin
Arm/Group | Usual Care | Active Treatment
Number analyzed (Participants) | 727 | 809
% glycolated hemoglobin
  Baseline | 8.92 (1.31) | 9.12 (1.48)
  6-Months: number analyzed (Participants) | 457 | 663
  6-Months | 8.26 (1.47) | 8.16 (1.37)
  12-Months: number analyzed (Participants) | 427 | 614
  12-Months | 8.15 (1.50) | 8.15 (1.40)

2. Secondary Outcome: Change in Systolic Blood Pressure (SBP)
Description: Systolic blood pressure (SBP) in each group will be assessed by the comparison of an average of the values obtained during routine outpatient clinical practice in 6-month windows preceding baseline and following the 6 and 12-month post-enrollment evaluation periods. In addition to measuring absolute values, the investigators will also examine the change in percentage of patients with an average SBP > 140.
Time Frame: 6 months and 12 months post-enrollment
Population: Only those with SBP values documented in the EHR during the evaluation windows were included in the number analyzed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Usual Care | Active Treatment
Number analyzed (Participants) | 727 | 809
mmHg
  Baseline: number analyzed (Participants) | 534 | 752
  Baseline | 139.6 (18.9) | 137.2 (17.5)
  6-Moths: number analyzed (Participants) | 555 | 721
  6-Moths | 139.6 (20.5) | 136.2 (18.7)
  12-Months: number analyzed (Participants) | 536 | 710
  12-Months | 139.3 (19.7) | 137.4 (19.5)

3. Secondary Outcome: Insulin Starts
Description: The number of participants who are not on insulin at baseline and are started on insulin during the 6 and 12-month post-enrollment periods will be totaled and compared for the SMA group and the no intervention control group. For the no intervention control group, baseline will be the date they are identified by the data manager. For the SMA group, baseline will be the date of the first SMA.
Time Frame: 6 months and 12 months post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Active Treatment
Number analyzed (Participants) | 727 | 809
Participants
  Baseline | 255 | 385
  6-Months | 247 | 418
  12-Months | 246 | 406

4. Secondary Outcome: Emergency Department (ED) Visits
Description: Major utilization events (admissions, bed days of care, and outpatient visits) will be collected from electronic medical records. Outpatient visits will be limited to those clinics most likely to be impacted by the intervention (e.g., primary care visits, diabetes specialty visits, and nurse visits).
Time Frame: 6 months and 12 months post-enrollment
Measure: Mean (Standard Deviation); unit: number of ED visits
Arm/Group | Usual Care | Active Treatment
Number analyzed (Participants) | 727 | 809
number of ED visits
  Baseline | 0.51 (1.24) | 0.54 (1.16)
  6-Months | 0.42 (1.04) | 0.68 (1.36)
  12-Months | 0.50 (1.26) | 0.60 (1.31)

5. Secondary Outcome: Statin Starts
Description: The number of participants who are not on a statin at baseline and are started on insulin during the 6 and 12-month post-enrollment periods will be totaled and compared for the SMA group and the no intervention control group. For the no intervention control group, baseline will be the date they are identified by the data manager. For the SMA group, baseline will be the date of the first SMA.
Time Frame: 6 months and 12 months post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Active Treatment
Number analyzed (Participants) | 727 | 809
Participants
  Baseline | 470 | 603
  6-Months | 456 | 617
  12-Months | 446 | 608

6. Secondary Outcome: Change in Number of Classes of Anti-hypertensive Meds
Description: Change in antihypertensive use (number of classes of prescribed anti-hypertensives) in each group will be assessed at baseline and following the 6 and 12-month post-enrollment evaluation periods. For the no intervention control group, baseline will be the date they are identified by the data manager. For the SMA group, baseline will be the date of the first SMA.
Time Frame: 6 months and 12 months post-enrollment
Population: Only those participants who were on at least one anti-hypertensive med during the evaluation windows were included in the number analyzed
Measure: Mean (Standard Deviation); unit: Number of classes of anti-hypertensives
Arm/Group | Usual Care | Active Treatment
Number analyzed (Participants) | 727 | 809
Number of classes of anti-hypertensives
  Baseline: number analyzed (Participants) | 548 | 655
  Baseline | 2.23 (1.27) | 2.38 (1.21)
  6-Months: number analyzed (Participants) | 517 | 668
  6-Months | 2.31 (1.28) | 2.38 (1.19)
  12-Months: number analyzed (Participants) | 513 | 660
  12-Months | 2.28 (1.19) | 2.39 (1.24)

7. Secondary Outcome: Change in Patient-reported Satisfaction With VA Care
Description: Patients' satisfaction with VA care will be assessed through surveys at baseline and 6 and 12 months post-enrollment for the SMA group. The following relates to the scale used:
  Scale name: VA Healthcare Satisfaction Scale Scale ranges: 1-6 (Strongly Disagree=1, Disagree=2, Slightly Disagree=3, Slightly Agree=4, Agree=5, Strongly Agree=6) Direction of range: Higher score indicates a better outcome
Time Frame: 6 months and 12 months post-enrollment
Population: Only those who completed each timepoint's survey and responded to the relevant scale items were included in the number analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Treatment
Number analyzed (Participants) | 448
units on a scale
  Baseline | 4.58 (1.04)
  6-Months: number analyzed (Participants) | 365
  6-Months | 4.97 (0.98)
  12-Months: number analyzed (Participants) | 345
  12-Months | 4.88 (1.08)

8. Secondary Outcome: Change in Patient-reported Diabetes Distress
Description: Patients' level of diabetes distress will be assessed through surveys at baseline and 6 and 12 months post-enrollment for the SMA group. The following relates to the scale used:
  Scale name: Diabetes Distress Scale Scale ranges: 1-5 (Not a Problem=1, Minor Problem=2, Moderate Problem=3, Somewhat Serious Problem=4, Serious Problem=5) Direction of range: Lower score indicates a better outcome
Time Frame: 6 months and 12 months post-enrollment
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Treatment
Number analyzed (Participants) | 451
units on a scale
  Baseline | 2.43 (1.02)
  6-Months: number analyzed (Participants) | 350
  6-Months | 2.19 (0.99)
  12-Months: number analyzed (Participants) | 315
  12-Months | 2.03 (0.93)

9. Secondary Outcome: Change in Patient-reported Degree of Diabetes Support
Description: Patients' degree of diabetes support will be assessed through surveys at baseline and 6 and 12 months post-enrollment for the SMA group. The following relates to the scale used:
  Scale name: Diabetes Support Scale Scale ranges: 1-6 (Strongly Disagree=1, Disagree=2, Slightly Disagree=3, Slightly Agree=4, Agree=5, Strongly Agree=6) Direction of range: Higher score indicates a better outcome
Time Frame: 6 months and 12 months post-enrollment
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Treatment
Number analyzed (Participants) | 446
units on a scale
  Baseline | 3.77 (1.30)
  6-Months: number analyzed (Participants) | 351
  6-Months | 4.29 (1.25)
  12-Months: number analyzed (Participants) | 314
  12-Months | 4.09 (1.37)

10. Secondary Outcome: Change in Patient-reported Degree of Self-Efficacy
Description: Patients' degree of self-efficacy will be assessed through surveys at baseline and 6 and 12 months post-enrollment for the SMA group. The following relates to the scale used:
  Scale name: Williams Self-Efficacy Scale Scale ranges: 1-6 (Strongly Disagree=1, Disagree=2, Slightly Disagree=3, Slightly Agree=4, Agree=5, Strongly Agree=6) Direction of range: Higher score indicates a better outcome
Time Frame: 6 months and 12 months post-enrollment
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Treatment
Number analyzed (Participants) | 449
units on a scale
  Baseline | 4.51 (1.05)
  6-Months: number analyzed (Participants) | 350
  6-Months | 4.84 (1.02)
  12-Months: number analyzed (Participants) | 312
  12-Months | 4.87 (1.05)

11. Secondary Outcome: Hospitalizations
Description: as for outcome 4
Time Frame: 6 months and 12 months post-enrollment
Measure: Mean (Standard Deviation); unit: number of hospitalizations
Arm/Group | Usual Care | Active Treatment
Number analyzed (Participants) | 727 | 809
number of hospitalizations
  Baseline | 0.12 (0.46) | 0.10 (0.36)
  6-Months | 0.12 (0.52) | 0.15 (0.56)
  12-Months | 0.14 (0.55) | 0.12 (0.52)

12. Secondary Outcome: Length of Hospitalizations
Description: as for outcome 4
Time Frame: 6 months and 12 months post-enrollment
Population: Only those participants who had at least one hospitalization during the evaluation windows were included in the number analyzed
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Care | Active Treatment
Number analyzed (Participants) | 727 | 810
days
  Baseline: number analyzed (Participants) | 61 | 71
  Baseline | 6.1 (12.7) | 3.1 (3.2)
  6-Months: number analyzed (Participants) | 56 | 84
  6-Months | 12.7 (33.2) | 6.3 (9.3)
  12-Months: number analyzed (Participants) | 63 | 64
  12-Months | 7.3 (9.2) | 8.6 (21.5)

13. Secondary Outcome: PCP Visits
Description: as for outcome 4
Time Frame: 6 months and 12 months post-enrollment
Measure: Mean (Standard Deviation); unit: number of PCP visits
Arm/Group | Usual Care | Active Treatment
Number analyzed (Participants) | 727 | 809
number of PCP visits
  Baseline | 1.65 (1.47) | 1.57 (1.30)
  6-Months | 1.04 (1.20) | 1.42 (1.37)
  12-Months | 1.11 (1.19) | 1.38 (1.29)

14. Secondary Outcome: Nurse Case Manager Visits
Description: as for outcome 4
Time Frame: 6 months and 12 months post-enrollment
Measure: Mean (Standard Deviation); unit: number of RNCM visits
Arm/Group | Usual Care | Active Treatment
Number analyzed (Participants) | 727 | 809
number of RNCM visits
  Baseline | 0.40 (1.12) | 0.42 (1.09)
  6-Months | 0.08 (0.38) | 0.29 (0.86)
  12-Months | 0.18 (0.74) | 0.23 (0.78)

15. Secondary Outcome: Endocrinology Visits
Description: as for outcome 4
Time Frame: 6 months and 12 months post-enrollment
Measure: Mean (Standard Deviation); unit: number of Endocrinology visits
Arm/Group | Usual Care | Active Treatment
Number analyzed (Participants) | 727 | 809
number of Endocrinology visits
  Baseline | 0.18 (0.69) | 0.21 (0.64)
  6-Months | 0.15 (0.68) | 0.20 (0.61)
  12-Months | 0.15 (0.62) | 0.21 (0.63)

ADVERSE EVENTS:
Time Frame: For each enrolled patient, adverse event data were collected from enrollment through 1 year 3 months post-enrollment.
Arm/Group | Usual Care | Active Treatment
All-Cause Mortality (participants affected / at risk) | 0/727 | 0/809
Serious Adverse Events (participants affected / at risk) | 0/727 | 0/809
Other Adverse Events (participants affected / at risk) | 0/727 | 0/809

LIMITATIONS AND CAVEATS:
1. Our study sites were VAs.
2. We did not collect survey data from the usual care group, so were unable to compare responses between the two arms.
3. All clinical outcomes were gathered from EHR data gathered through clinical visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT02132676/Prot_SAP_000.pdf